CLINICAL TRIAL: NCT01268787
Title: A Phase I, Randomized, Open-Label Study to Evaluate the Safety and Immunogenicity of EV71 Vaccine Administrated With Adjuvant AlPO4 in Health Volunteers
Brief Title: A Study to Evaluate the Safety and Immunogenicity of EV71 Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QCR-10013
Record Dates: First submitted 2010-12-30; First posted 2010-12-31 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2013-10

CONDITIONS: Enterovirus Infection
MeSH Terms: conditions — Enterovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EV 71 vaccine 5ug (Active Comparator): EV71 Vaccine 5ug
  Interventions: Biological: EV71 vaccine
- EV 71 vaccine 10ug (Experimental): EV71 vaccine 10ug
  Interventions: Biological: EV71 vaccine

INTERVENTIONS:
Biological: EV71 vaccine — Two-vaccination 0.25ml or 0.5ml dose assigned to two groups.
  Other Names: EV71 vac

SUMMARY:
This study is aims to evaluate the safety, reactogenicity and immunogenicity of EV71 vaccine at a 0.25ml or 0.5ml dose in health volunteers

DETAILED DESCRIPTION:
This is a phase I, prospective, randomized, open-label, two-center study. A total 60 healthy volunteers will be screened for baseline characteristic inclusion/exclusion criteria after providing a written informed consent. Eligible subjects will be recruited and equally randomized to either receive 2 doses of EV71 vaccine 0.25ml or 0.5ml. All subjects should be followed till Day 210.

ELIGIBILITY:
Inclusion Criteria:

* Subject who is free of obvious health problems
* Able and willing to comply with the study procedure adn give written informed consent

Exclusion Criteria:

* Female who is pregnant/lactating or planning to be pregnant
* Body mass index(BMI) > 35
* Oral temperature > 37.5 Celsius at the time of planned vaccination
* Subject with any abnormal laboratory results at screening
* With a history of herpangina, hand-foot-mouth disease, acute hemorrhagic conjunctivitis or acute gastrointestinal illness associated with enterovirus infection in the past 3 months
* Has been diagnosed with neurological, pulmonary, cardiovascular, hematological, hepatic or renal disorder
* With a history of hypersensitivity to vaccine or allergic disease
* Use of any investigational/non-registered product within 30 days prior to vaccination
* Use of immunoglobulins or any blood products within 3 months prior to vaccination
* Chronic administration of immunosuppressants or other immunomodulators within 5 months prior to vaccination

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-12; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Primary endpoint | 210 Days
  The percentage, intensity and relationship to vaccination of local and systemic signs and symptoms at a 0.25ml and 0.5ml dose

CONTACTS AND LOCATIONS:
Overall Officials: Pele Chong, Ph.D., Study Chair — National Health Research Institutes, Taiwan; Chia-Chyi Liu, Ph.D., Study Director — National Health Research Institutes, Taiwan; C P Fung, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan; S M Hsieh, M.D, Principal Investigator — Taipei Meidcal College
Locations (2):
- Taiwan (2):
  - Taipei Veterans General Hospital, Taipei, Shihlin District
  - National Taiwan University Hospital, Taipei, Zhongshan Distric

REFERENCES:
- [Derived] Chou AH, Liu CC, Chang JY, Jiang R, Hsieh YC, Tsao A, Wu CL, Huang JL, Fung CP, Hsieh SM, Wang YF, Wang JR, Hu MH, Chiang JR, Su IJ, Chong PC. Formalin-inactivated EV71 vaccine candidate induced cross-neutralizing antibody against subgenotypes B1, B4, B5 and C4A in adult volunteers. PLoS One. 2013 Nov 21;8(11):e79783. doi: 10.1371/journal.pone.0079783. eCollection 2013. PMID 24278177
- [Derived] Cheng A, Fung CP, Liu CC, Lin YT, Tsai HY, Chang SC, Chou AH, Chang JY, Jiang RH, Hsieh YC, Su IJ, Chong PC, Hsieh SM. A Phase I, randomized, open-label study to evaluate the safety and immunogenicity of an enterovirus 71 vaccine. Vaccine. 2013 May 7;31(20):2471-6. doi: 10.1016/j.vaccine.2013.03.015. Epub 2013 Mar 27. PMID 23541623